CLINICAL TRIAL: NCT01690598
Title: Veliparib (ABT888) and Topotecan (Hycamtin®) for Patients With Platinum-Resistant or Partially Platinum-Sensitive Relapse of Epithelial Ovarian Cancer With Negative or Unknown BRCA Status
Brief Title: Veliparib and Topotecan for Relapsed Ovarian Cancer With Negative or Unknown BRCA Status
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VeTo
Record Dates: First submitted 2012-09-17; First posted 2012-09-24 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Ovarian Cancer
Keywords: Epithelial ovarian cancer; BRCA mutation; Platinum resistant; Platinum sensitive; Relapsed ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — veliparib; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Veliparib and Topotecan (Experimental)
  Interventions: Drug: Veliparib; Drug: Topotecan

INTERVENTIONS:
Drug: Veliparib — Veliparib (tablet) twice daily on days 1-3, 7-9, and 14-16 in a 28 days cycle. In phase I the starting dose is 30 mg x 2.
Drug: Topotecan — 2 mg/m² iv over 30 minutes on days 2, 8, and 15 in cycles of 28 days. Topotecan is dosed at a maximum body surface area of 2 m².

SUMMARY:
The purpose of this study is to investigate the effect of combined topotecan and veliparib (ABT888) treatment in relapsed ovarian cancer with tumor progression and negative or unknown BRCA mutation status.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed epithelial, primary fallopian or primary peritoneal cancer.
2. Verified progression by either RECIST criteria and/or GCIG CA125 criteria after previous first line chemotherapy or progression after later lines of cytotoxic treatment.
3. Platinum resistance or partially platinum sensitive disease

   * Relapsed within six months of prior first line/later lines of platinum-based therapy or
   * Relapsed within six-twelve months of prior first line/later lines of platinum-based therapy
4. Age ≥ 18 years.
5. Performance status 0-2.
6. Measurable disease by RECIST 1.1 or CA125 GCIG criteria
7. Adequate bone marrow function, liver function, renal function and coagulation parameters (within 7 days prior to enrollment):

   * WBC ≥ 3.0 x 10^9/l or neutrophils (ANC) ≥ 1.5 x 10^9/l
   * Platelet count ≥ 100 x 109/l
   * Hemoglobin ≥ 9.7 g/dl (6 mmol/L)
   * Serum bilirubin ≤ 1.5 x ULN
   * Serum transaminases ≤ 2.5 x ULN
   * Serum creatinine ≤ 1.5 x ULN
8. Written informed consent.
9. Tissue available for BRCAness analysis/BRCA mutation analysis.

Exclusion Criteria:

1. Prior treatment with a PARP inhibitor.
2. Patients with BRCA1/2 germline mutation.
3. Platinum-refractory disease (disease that progressed or was stable during prior platinum therapy)
4. Patients who have received (or are planning to receive) treatment with any other investigational agent, or who have participated in another clinical trial within 28 days prior to entering this trial.
5. Pregnant or breast-feeding. For fertile women a negative pregnancy test at screening is mandatory.
6. Fertile patients not willing to use acceptable and safe methods of contraception during and for 6 months after treatment
7. Other present or previous malignancy except curatively treated cervical cancer stage I, non-melanotic skin cancer or other cancer with minimal risk of relapse. Previous breast cancer is allowed, if disease free follow-up at least five years prior to enrollment.
8. CNS metastasis.
9. History of any chronic medical or psychiatric condition or laboratory abnormality, which is not medically controlled or in the opinion of the Investigator may increase the risks associated with study drug administration (e.g. diabetes, cardiac diseases, hypertension, renal or liver disease).
10. Allergy to the ingredients of the study medication.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-11; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Phase I: Maximum tolerated dose, dose limiting toxicity and thus recommend phase II dose of veliparib | 1 month
Phase II: To investigate response rates (based on either CA125 GCIG or RECIST criteria) of combination topotecan and veliparib (ABT888) in relapsed ovarian cancer with negative or unknown BRCA status | Every three months, up to 3 years

SECONDARY OUTCOMES:
Progression free survival of ovarian cancer patients treated with topotecan and veliparib | Every three months up to three years
Overall survival of ovarian cancer patients treated with topotecan and veliparib | Every three months, up to three years

CONTACTS AND LOCATIONS:
Overall Officials: Anders Jakobsen, MD, DMSc, Study Chair — Vejle Hospital; Hanne Kanstrup, MD, Principal Investigator — Vejle Hospital
Locations (1):
- Department of Oncology, Vejle Hospital, Vejle, Denmark

REFERENCES:
- [Derived] Hjortkjaer M, Kanstrup H, Jakobsen A, Steffensen KD. Veliparib and topotecan for patients with platinum-resistant or partially platinum-sensitive relapse of epithelial ovarian cancer with BRCA negative or unknown BRCA status. Cancer Treat Res Commun. 2018;14:7-12. doi: 10.1016/j.ctarc.2017.09.001. Epub 2017 Sep 27. No abstract available. PMID 30104007